CLINICAL TRIAL: NCT04516109
Title: Modifications of Devices for Hip Arthroscopy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 19-2755
Record Dates: First submitted 2020-07-08; First posted 2020-08-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hip Arthroscopy
Keywords: Hip arthroscopy; Arthroscopy; Labral repair; bone grafting; Total hip arthroplasty

STUDY DESIGN:
Intervention Model Description: All eligible patients undergoing hip arthroscopy by the principal investigator will be assigned to one of two groups for analysis, based on the appropriate SOC surgical treatment for FAI, hip dysplasia, or a combination of the two. All patients will undergo hip arthoscopy with the use of the modified hip capsule slotted cannula.
Who Masked: Investigator
Masking Description: We will be utilizing anonymous staff surveys. After the staff within the operating room (scrub, circulator, PA, and fellow) completes the paper survey (following the procedure), the staff member (who did not use the device per specific surgery) will administer the survey and seal in an envelope, which will be sent to the PRA. Thus, these responses will be blinded to the PI.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthrosocpic labral repair (Active Comparator): Patients undergoing arthroscopic labral repair with the use of the modified hip capsule slotted cannula.
  Interventions: Device: Modified hip capsule side fixed slotted cannula
- Arthroscopic bone grafting (Active Comparator): Patients undergoing arthroscopic bone grafting of subchrondral cyst with the use of the modified bone graft delivery tool set and modified hip capsule slotted cannula.
  Interventions: Device: Modified hip capsule side fixed slotted cannula; Device: Modified bone graft delivery tool set

INTERVENTIONS:
Device: Modified hip capsule side fixed slotted cannula — Modified hip capsule side fixed slotted cannula used during surgery to allow for continued access to the hip joint.
Device: Modified bone graft delivery tool set — Modified bone graft delivery tool set for grafting subchrondral cysts arthroscopically during hip arthroscopy procedure.
  Arms: Arthroscopic bone grafting

SUMMARY:
This is protocol is intended to demonstrate the principal investigator's improvements and modifications of a hip capsule side fixed slotted cannula for continued access to the hip joint and a bone graft delivery tool set for grafting subchrondral cysts during hip arthroscopy procedure.

DETAILED DESCRIPTION:
Femoroacetabular impingement (FAI) and acetabular dysplasia represent the two most common causes of secondary osteoarthritis of the hip1-3 and the two main indications for Hip Preservation procedures. Most patients with these pathologies will undergo Hip Arthroscopy, either alone, or combined with bony realignment procedures. Hip arthroscopy has grown exponentially over the past 15 years and is currently being leveraged in the diagnosis and treatment of a wide range of hip joint problems.

In an effort to improve surgical techniques, make surgeries faster and reproducible, mitigate complications and increase patient safety, surgeons modify and improve commercially available and commonly used non-significant risk devices with the above goals in mind.

For these reasons, the Principal Investigator (PI) modified and improved two devices for hip arthroscopy. These include the modified (1) hip capsule side fixed slotted cannula for continued access to the hip joint and (2) bone graft delivery tool set for grafting subchrondral cysts arthroscopically during hip arthroscopy procedure. After utilizing these modified devices clinically, the PI has been impressed with their impact and thus aims to demonstrate that the modifications provide significant improvements in surgical flow and technique, minimize surgical time (per technical phase), minimize surgical costs, result in an absolute low incidence of surgical complications, and ultimately improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 60 years diagnosed with FAI, Hip Dysplasia or the combination of the two.
* Persistent hip pain accompanied by mechanical symptoms refractory to nonoperative management lasting at least 3 months.
* Reproducible clinical examination findings suggestive of impingement and/or decreased range of motion, and positive radiographic findings on radiography, computed tomography with 3-dimensional reconstruction, and magnetic resonance imaging.
* Joint-space width > 3 mm on all views of plain radiography and 3-dimensional computed tomography.
* Patients undergoing hip arthroscopy for the treatment of FAI, Hip Dysplasia, or the combination of the two by the Principal Invesitgator.

Exclusion Criteria:

* Age <18 years.
* Prisoners.
* Pregnant women.
* Decisionally challenged.
* Does not speak or understand English.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Surgical time per technical phase measured in minutes | 1 Day
  * We aim to demonstrate that the use of the modified device for hip arthroscopy is fast and efficient as measured by surgical time per technical phase (i.e. arthroscopic labral repair phase and arthroscopic bone grafting phase).
  * Arthroscopic Labral Repair Phase: During hip arthoscopy, the surgical time of the arthroscopic labral repair phase will be collected.
  * Arthroscopic Bone Grafting Phase: During hip arthoscopy, the surgical time of the bone grafting of the hip joint phase will be collected.
  * In this design, the technical phase recorded will either be: 1) duration of arthroscopic labral repair phase (in patients only undergoing arthroscopic labral repair) or 2) duration of arthroscopic bone grafting phase (in patients undergoing arthroscopic bone grafting).

SECONDARY OUTCOMES:
Rate of Surgical Complications | Up to 24 months
  Total number of complications determined to be related to the hip arthroscopy procedure.
Surgical costs per device used | 1 Day
  Cost to use each device in surgery, measured in US dollars.
Patient Outcomes: Post-operative Pain | Post operative up to Day 9
  Pain, as assessed via a visual analog scale. Possible scores range from 0-100, with 0 indicating no pain and 100 indicating the most severe pain and a worse outcome.
Patient Outcomes: Change in Pain | Pre-treatment, Week 6, Month 3, Month 6, Month 12, Month 24
  Pain, as assessed via a visual analog scale. Possible scores range from 0-100, with 0 indicating no pain and 100 indicating the most severe pain and a worse outcome.
Patient Outcomes: Change in International Hip Outcome Tool (IHOT-12) Scores | Pre-treatment, Week 6, Month 3, Month 6, Month 12, Month 24
  The International Hip Outcome Tool (IHOT-12) measures both health-related quality of life and changes after treatment in young, active patients with hip disorders. Patients indicate their responses to the various questions by marking a 100 mm visual analog scale. The total score is calculated by calculating the mean of the participant's responses. Possible scores range from 0-100 with 0 indicating the worst and 100 indicating the best possible quality of life.
Patient Outcomes: Change in Non-Arthritic Hip Scores | Pre-treatment, Week 6, Month 3, Month 6, Month 12, Month 24
  The Non-Arthritic Hip score is a self-administered hip score measuring function and quality of life designed for use in younger patients with higher activity demands and treatment expectations than older patients with degenerative joint disease. Possible scores range from 0-4, with 0 indicating the worst and 4 indicating the best level of function and outcome for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei-Dan, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado, Hip Preservation Center, Orthopedic Department, Boulder, Colorado
  - UCHealth Steadman Hawkins Clinic - Denver, Englewood, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beck M, Kalhor M, Leunig M, Ganz R. Hip morphology influences the pattern of damage to the acetabular cartilage: femoroacetabular impingement as a cause of early osteoarthritis of the hip. J Bone Joint Surg Br. 2005 Jul;87(7):1012-8. doi: 10.1302/0301-620X.87B7.15203. PMID 15972923
- [Background] Zhang C, Li L, Forster BB, Kopec JA, Ratzlaff C, Halai L, Cibere J, Esdaile JM. Femoroacetabular impingement and osteoarthritis of the hip. Can Fam Physician. 2015 Dec;61(12):1055-60. PMID 26668284
- [Background] Lung R, O'Brien J, Grebenyuk J, Forster BB, De Vera M, Kopec J, Ratzlaff C, Garbuz D, Prlic H, Esdaile JM. The prevalence of radiographic femoroacetabular impingement in younger individuals undergoing total hip replacement for osteoarthritis. Clin Rheumatol. 2012 Aug;31(8):1239-42. doi: 10.1007/s10067-012-1981-9. Epub 2012 May 3. PMID 22552857
- [Background] Huo MH, Parvizi J, Bal BS, Mont MA; Council of Musculoskeletal Specialty Societies (COMSS) of the American Academy of Orthopaedic Surgeons. What's new in total hip arthroplasty. J Bone Joint Surg Am. 2008 Sep;90(9):2043-55. doi: 10.2106/JBJS.H.00741. No abstract available. PMID 18762667
- [Background] Kelly BT, Williams RJ 3rd, Philippon MJ. Hip arthroscopy: current indications, treatment options, and management issues. Am J Sports Med. 2003 Nov-Dec;31(6):1020-37. doi: 10.1177/03635465030310060701. PMID 14623676
- [Background] Philippon MJ, Stubbs AJ, Schenker ML, Maxwell RB, Ganz R, Leunig M. Arthroscopic management of femoroacetabular impingement: osteoplasty technique and literature review. Am J Sports Med. 2007 Sep;35(9):1571-80. doi: 10.1177/0363546507300258. Epub 2007 Apr 9. PMID 17420508
- [Background] Huo MH, Parvizi J, Bal BS, Mont MA. What's new in total hip arthroplasty. J Bone Joint Surg Am. 2009 Oct;91(10):2522-34. doi: 10.2106/JBJS.I.00801. No abstract available. PMID 19797590
- [Background] Leunig M, Werlen S, Ungersbock A, Ito K, Ganz R. Evaluation of the acetabular labrum by MR arthrography. J Bone Joint Surg Br. 1997 Mar;79(2):230-4. doi: 10.1302/0301-620x.79b2.7288. PMID 9119848
- [Background] Tsai SW, Chen CF, Wu PK, Chen TH, Liu CL, Chen WM. Modified anterolateral approach in minimally invasive total hip arthroplasty. Hip Int. 2015 May-Jun;25(3):245-50. doi: 10.5301/hipint.5000218. Epub 2015 Feb 12. PMID 25684250
- [Background] Wang Y, Xu H, Ding M, Zhen Z, Lu Q, Liao B, Shangguan L. Permanently Avoiding Steam on Camera for Arthroscopy by a Simple Device. Arthrosc Tech. 2018 Dec 17;8(1):e47-e49. doi: 10.1016/j.eats.2018.08.029. eCollection 2019 Jan. PMID 30899650
- [Background] RStudio: Integrated Development for R. [computer program]. Version 1.1.456. Boston, MA: RStudio, Inc.; 2016